CLINICAL TRIAL: NCT04296734
Title: Effects of a Prenatal Depression Preventive Intervention on Parenting and Young Children's Self-Regulation and Functioning (EPIC)
Brief Title: Prenatal Depression Prevention Effects on Parenting and Young Child Self-Regulation and Functioning
Acronym: EPIC
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Darius Tandon, Associate Professor, Department of Medical Social Sciences Co-Director, Center for Community Health, Northwestern University
Other Study IDs: HD097215; GRANT12740559 (Other Grant/Funding Number: NICHD); 1R01HD097215-01A1 (NIH)
Record Dates: First submitted 2019-11-13; First posted 2020-03-05 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Postpartum Depression; Child Development; Parenting; Child Self-Regulation
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Mothers and Babies — Mothers & Babies (MB) is a program that promotes healthy mood management by teaching pregnant women and new moms how to effectively respond to stress in their lives through increasing the frequency of thoughts and behaviors that lead to positive mood states. Designed as a perinatal depression prevention, the Mothers & Babies targets three specific risk factors: limited social support, lack of pleasant activities, and harmful thought patterns.

SUMMARY:
Poor parenting practices and compromised child self-regulation when a child is 2 ½ - 4 ½ years old are foundational in promoting their later healthy development and adaptive functioning. This project will test whether targeting depressive symptoms with a prenatal preventive intervention prevents disruptions in well-regulated parenting and child self-regulation known to affect families with depressed mothers. This project may have great benefit to society, as preventive interventions delivered prenatally have the potential to influence long-term trajectories of parenting practices and child development which, in turn, can chart a course for future child health and well-being.

DETAILED DESCRIPTION:
The proposed R01 project Effects of a Prenatal Depression Preventive Intervention on Parenting and Young Children's Self-Regulation and Functioning (EPIC) examines whether a prenatal depression prevention intervention-Mothers and Babies (MB)-improves parenting practices and child self-regulation through 54 months of age. The investigators build on an existing cluster randomized controlled trial that enrolled 874 diverse, low-income women from 36 home visiting (HV) programs. The investigators anticipate 598 of these women will be eligible for EPIC (489 intervention, 109 control) and the research team will enroll an additional 260 control participants as part of this R01, for a total sample of 858. The research team will also enroll 429 fathers. Perinatal depression is consistently linked to poor parenting practices and poor child self-regulation. This project builds on previous work that has demonstrated MB's effects on improving maternal mental health outcomes and will examine the intervention's longer-term impact on parenting and child self-regulation from 30-54 months of age. Intervention participants will have received the six-week MB intervention delivered in a group format in addition to usual HV services while control participants will have only received HV services. Data collection for the R01 includes maternal self-report with all 858 participants every six months, beginning at 30 months postpartum and continuing until 54 months postpartum. An intensive sub-study of parenting and child development will occur at 36, 42, and 48 months for a subset of 460 participants (230 intervention, 230 control). Paternal self-report surveys will occur at 30, 42, and 54 months. There are three specific aims. First, the investigators test the hypothesis that MB improves parenting and child self-regulatory skill acquisition through 54 months of age. The investigators will use intent-to-treat as well as propensity score adjusted analysis. Second, the investigators test hypotheses about the maternal mechanisms by which MB influences parenting and child self-regulation. The investigators hypothesize that MB intervention effects will be mediated by core skills targeted by MB-in particular, increased awareness of thoughts and feelings and increases in mood regulation-as these cognitive-behavioral skills are deficient in mothers with depressive symptoms and compromise mothers' ability to engage in parenting practices that promote young children's self-regulation. Third, the investigators will examine fathers' and other key sociodemographic variables' role in moderating the impact of MB on mother's parenting and the child's self-regulation. The public health significance and innovation of this project is substantial. Addressing maternal mental health has been identified as a highly impactful enhancement to HV programs. If, as expected, the investigators are able to generate a robust science base that precisely identifies mechanisms and outcomes impacted by the intervention in young children among our racially and ethnically diverse sample, HV programs currently using MB are likely to enhance their programmatic outcomes. Moreover, given the large number of HV programs that could adopt MB nationally, findings from this study can provide powerful data suggesting that MB become integrated into their core set of services.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

Women enrolled in parent-study:

* ≥ 16 years of age
* ≤33 weeks' gestation upon referral
* English or Spanish speaking

New Cohort:

* English or Spanish speaking
* ≥ 18 years of age
* Have a child 18-30 months old at the time of recruitment

Partners of female study participants:

* ≥ 18 years of age
* English or Spanish speaking
* Have contact with the child of one of the existing/new female participants

Min Age: 18 Months | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This study builds on a currently ongoing parent study that enrolled pregnant women from home visiting (HV) programs across seven states to examine the effects of a cognitive-behavioral therapy (CBT) intervention-Mothers and Babies (MB)-on maternal mental health through six months postpartum. This follow-up study will retain the same cohort of women enrolled in that study and recruit additional women to serve as control participants. Children will be ages 30 months to 54 months in this study. The research team will also recruit a cohort of fathers in this follow-up study
Sampling Method: Non-Probability Sample
Enrollment: 960 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Maternal depressive symptoms | Child age 30-54 months
  Measured by the 16-item Quick Inventory of Depressive Symptomatology (QIDS). Total score ranges from 0-27. Scores between 0-5 (no depression); 6-10 (Mild Depression); 11-15 (Moderate); 16-20 ( Severe); 21+ (Very Severe) .
Parenting outcomes ) of parenting self-efficacy (SE) and Parenting Hostile Reactive Behavior (HRB) | Child age 30-54 months
  Measured by the Parental Cognitions and Conduct Toward the Infant Scale (PACOTIS). Scores range from 0-10. Higher mean scores indicate greater self-efficacy, hostile-reactive parenting, perceived parental impact, and parental overprotection
Child self-regulation outcomes | Child age 30-54 months
  Measured by the Early Childhood Behavior Questionnaire-Very Short Form (ECBQ-VS). Items indicated with an R on the items-by-scale list below are reverse-scored. Sum the scores for items receiving a numerical response.
  Negative Affect (12 items): 16,17,19,32,2,26,10,22,23,1,33,34R Surgency (12 items): 4,13,18,20,24,6,11,9,25,3,30,36 Effortful Control (12 items): 21,27,31,8,15,35,7,14R,12R,29,5,28
  Effortful Control measured by the Multidimensional Assessment Profile of Disruptive Behavior Short Form (MAP-DB) Temper Loss Subscale. A sum of the 49 short-form items to indicate total Disruptive Behavior (DB); A sum of the 22 TL items (15+7) to indicate Temper Loss. The scale goes from 0 (never) to 5 (many times each day). Higher scores indicate higher levels of problems.

SECONDARY OUTCOMES:
Maternal mental health and cognitive-behavioral skills | Child age 30-54 months
  1. Behavioral activation measured by the Behavioral Activation for Depression Scale (BADS). The BADS consists of 25 items, each rated on a 7-point scale, with higher scores indicating greater behavioral activation.
  2. Decentering measured by Experiences Questionnaire (EQ). Total Score is the sum of all 20 items. The higher the score the higher the decentering/rumination.
  3. Social support measured by Medical Outcomes Study Social Support Survey (MOS-SS). 19 items, with greater scores indicating more perceived social support.
  4. Perceived stress measured by the 4-item Perceived Stress Scale (PSS-4). Higher scores are correlated to more stress.
  5. Relationship with partner measured by the Revised Dyadic Adjustment Scale (RDAS). The total score is the sum of the responses to the 7 items. Higher scores indicate greater relationship satisfaction.
Parenting outcomes of parental positive affect, sensitive responsiveness, and verbalizations | Child age 36-48 months
  Measured by the Brief Early Relational Assessment (BERA). Coding factors are Child, Parent, and Dyadic. Each item on a factor is scored from 1-5 with 1-2=no concern, 3=some concern, 4-5=areas of strength. All items on a factor are added and divided by the number of items on the factor to get a mean score. There is no overall score.
Child self-regulation outcomes | Child age 36-48 months
  Measured by: a. Devereaux Early Childhood Assessment (DECA) Initiative, Attachment/relationships, Self-regulations subscales (Time frame: Child age 30-54 months). Four subscales: initiative, self-regulation, attachment/relationships, behavioral concerns. Each item rated 0-4. For each subscale, sum responses to get a scale raw score. Use the scoring guide to get the child's Protective Factor Profile based on the Self-regulation, attachment/relationships, and behavioral concerns raw scores.
  b. Disruptive Diagnostic Observation Schedule (DB-DOS) Problems in Behavioral Regulation. 3 domains: Problems in anger modulation, problems in behavioral regulation, competence. Ratings are made on a 4-point scale ranging from 0 (none) to 3 (high). Scores are derived as sums of each domain.

CONTACTS AND LOCATIONS:
Overall Officials: S. Darius Tandon, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diebold A, Johnson JK, Brennan M, Ciolino JD, Petitclerc A, Wakschlag LS, Garfield CF, Yeh C, Lovejoy A, Zakieh D, Tandon SD. Testing the effects of a prenatal depression preventive intervention on parenting and young children's self-regulation and functioning (EPIC): protocol for a longitudinal observational study. BMC Public Health. 2021 Jul 10;21(1):1368. doi: 10.1186/s12889-021-11385-5. PMID 34246233